CLINICAL TRIAL: NCT05590845
Title: Evaluating Patient Knowledge About Perioperative Neurocognitive Disorders (KNOW-PND Study)
Status: Recruiting | Type: Observational
Sponsor: Université Libre de Bruxelles (Other)
Responsible Party: Principal Investigator, Sarah Saxena, PI, Université Libre de Bruxelles
Other Study IDs: Know-PND
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-05

CONDITIONS: Anesthesia Complication
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Survey — Patients, 65 and above, scheduled for elective total hip replacement surgery, will be invited to participate in a survey (consisting of 15 questions) testing their knowledge regarding PND.
  After completion of the survey, patients will receive a standard preoperative brochure on anaesthesia-related topics and delirium.
  T-MOCA scores will be collected (22 = perfect score; <18 = cutoff for cognitive impairment) (through a pre-operative telephone call).
  Six weeks post-operatively patients will once again be called for T-moca scores.
  Initially a feasibility study for 1/3 of sample size will be done.

SUMMARY:
Neurocognitive disorders remain one of the major perioperative complications. They are associated with delayed recovery, prolonged length of hospital stay and impacts on patients' quality of life. The incidence of PND ranges from 15-50%.

While several causes have been investigated, PND seems to be due to the non-resolution of an inflammatory cascade, making some patients more at risk than others. As such, major risk factors include old age and lower education levels.

As the global proportion of people aged 60 and above between 2015 and 2050 will increase from 12% to 22% and worldwide surgeries increases to >300 million procedures per annum the incidence of perioperative neurocognitive disorders with high morbidity and mortality will go up.

In 2015, the American Society of Anesthesiologists (ASA) launched the 'Perioperative Brain Health Initiative' to increase awareness about perioperative neurocognitive disorders. (PND) While physicians seems to be more and more aware about this condition, data regarding patient awareness are not available.

An observational, single-centre, cross-sectional survey study (with initially a feasibility study) will be conducted in patients, 65 years and above undergoing elective total hip replacement surgery at AZ Sint-Jan (Brugge, Belgium) to assess patients' basic knowledge regarding PND.

ELIGIBILITY:
Inclusion Criteria:

* age 65 and above
* ASA score 1 to 3
* scheduled for elective hip surgery.

Exclusion Criteria:

* insufficient knowledge of Dutch
* known neuropsychiatric conditions

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients scheduled for elective total hip replacement surgery.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
PND knowledge | 1 week pre-operatively
  Patient knowledge regarding PND will be evaluated through 15 yes/no questions

SECONDARY OUTCOMES:
Baseline cognition | 1 week pre-operatively
  Baseline T-moca scores will be documented in order to evaluate PND presence.
PND | 6 weeks post-operatively
  T-moca scores will be documented post-operatively (and compared to baseline scores) in order to evaluate PND presence.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Saxena, MD;PHD, Principal Investigator — AZ Sint-Lucas Brugge
Locations (1):
- AZ Sint-Jan Brugge Oostende AV, Bruges, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request, anonymous data will be shared.